CLINICAL TRIAL: NCT03729336
Title: Midstream Urine Collection Device Compared to Catheterized Sample: Contamination and Patient Satisfaction.
Brief Title: PEEZY Midstream Urine Device Compared to Catheterized Urine Sample
Acronym: PEEZY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Forte Medical (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 018-702
Record Dates: First submitted 2018-10-26; First posted 2018-11-02 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-02

CONDITIONS: Lower Urinary Tract Symptoms; Lower Urinary Tract Infection
Keywords: urine specimen; contamination
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Catheters; Urine Specimen Collection

STUDY DESIGN:
Intervention Model Description: Patient spontaneously voids in the bathroom using PEEZY (research sample). Within 10 minutes, patient is catheterized during physical exam (control sample) for post-void residual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEEZY specimen (Experimental): All subjects will use PEEZY to give a urine specimen.
  Interventions: Device: Midstream urine collection device
- CATHETER specimen (Placebo Comparator): All subjects will use CATHETER (performed by their clinician) to give a urine specimen, following PEEZY use.
  Interventions: Device: Catheter for urine collection

INTERVENTIONS:
Device: Midstream urine collection device — Non-invasive midstream urine collection device
  Other Names: PEEZY
  Arms: PEEZY specimen
Device: Catheter for urine collection — In-and-out catheter obtains urine through the urethra.
  Other Names: Straight catheter
  Arms: CATHETER specimen

SUMMARY:
Urine culture and microscopic urinalysis will be compared between 2 collection methods: PEEZY midstream urine collection, and urethral catheter collection.

DETAILED DESCRIPTION:
Female patients presenting to the Baylor Scott & White Health (Temple, TX) Urology clinic for complaints of lower urinary tract symptoms will be included. They will be approached by a clinical research coordinator and given more information. If they meet eligibility by screening, consents will be completed.

Patients will proceed with their regular clinic visit with their clinician. Just prior to the physical exam, patients will use the PEEZY device to give a urine specimen in the privacy of the bathroom. The package with PEEZY includes the simple instructions for use. Patients return to the clinic room and the physical exam proceeds. An in-and-out catheter is used to obtain a post-void residual as well as a control urine specimen. After the remainder of the patient routine exam is complete, they will fill out a brief questionnaire.

The 2 specimens will then be delivered to the lab. The clinical research coordinator will store consents and questionnaires that include the subjects study identification number in individual opaque envelopes that will be kept in a locked drawer accessible to only the investigators.

ELIGIBILITY:
Inclusion Criteria:

* Females presenting to the Urology or Urogynecology clinic for consultation or evaluation of lower urinary tract complaints.

Exclusion Criteria:

* Known pregnancy
* Use of antimicrobial oral or vaginal therapy in the past 4 weeks
* Use of Pyridium in the past 4 weeks

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Contamination of urine specimen with urethral and vaginal flora | 2 specimens from each subject (1 from each arm) will be taken to the lab for urinalysis and culture immediately after specimens are given. Culture results will be reported in 48 hours. After results are recorded, no further assessment of this outcome.
  Contamination defined as: presence of urethral or vaginal flora on urine culture OR epithelial cell presence in urinalysis

SECONDARY OUTCOMES:
Visual Analog Scale (this is the only title for this scale) | Performed one time immediately after intervention. This will not be repeated.
  On a questionnaire: patient rates level of distress experienced during each urine donation method. The scale is from 1 to 10. On this scale 10 is associated with the word "agonizing", 8 is associated with "horrible", 4 is associated with "uncomfortable", 2 is associated with "annoying", and 0 is associated with "None". Unbearable distress is marked near 10. No distress is marked near 0. On this scale responses can only be reported as a number from 0-10, and a lower number indicates a better outcome. There are no subscales.

OTHER OUTCOMES:
Patient Preference | Performed one time immediately after intervention. This will not be repeated.
  Questionnaire created by investigator asks: Which way would you prefer to give a urine sample, if needed in the future? PEEZY or catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel High, DO, Principal Investigator — Baylor Scott and White Health
Locations (1):
- Baylor Scott and White Health, Temple, Texas, United States

IPD SHARING:
Plan to Share IPD: No